CLINICAL TRIAL: NCT07181668
Title: Perioperative Low-Level Light Therapy for Ocular Surface Protection in Patients Undergoing Femto-LASIK: A Prospective Double-masked, Randomized Controlled Study
Brief Title: Effect of Low-Level Light Therapy on Ocular Surface Parameters in Patients Undergoing Femto-Lasik Surgery
Acronym: LLLT-Lasik
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Timofte Zorila Mihaela Madalina, Principal investigator, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Grigore T. Popa n.54/29.07.24
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction (Disorder); Ocular Surface Disease
Keywords: Dry eye disease; LLLT; Photobiomodulation
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, double-masked, parallel-group trial. Eligible participants undergoing femtosecond laser-assisted in situ keratomileusis (Femto-LASIK) are randomly assigned in a 1:1 ratio to receive either low-level light therapy (LLLT) or a sham treatment. Interventions are administered perioperatively (1 week before and 1 week after surgery), and all clinical outcomes are assessed at baseline, 1 week, 1 month, and 3 months postoperatively. Participants remain in their assigned group for the duration of the study, with no crossover between groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLLT Group (Experimental): Participants in the LLLT group received periocular low-level light therapy (LLLT) using the Eye-light® device (Espansione Marketing S.p.A., Italy) for 15 minutes per session, one week before and one week after femtosecond laser-assisted in situ keratomileusis (Femto-LASIK). The device delivers red light at 633 ± 10 nm through closed eyelids, targeting the periocular region and meibomian glands to support tear film stability and reduce ocular discomfort. All participants underwent standard Femto-LASIK surgery and received identical postoperative care, including topical antibiotics, corticosteroids, and preservative-free artificial tears. Of the 31 patients initially assigned to the LLLT group, 6 were lost to follow-up, leaving 23 patients (46 eyes) for the final analysis.
  Interventions: Device: Low-Level Light Therapy
- Sham Group (Sham Comparator): Participants in the Control group underwent a sham treatment using the same Eye-light® device with minimal energy (<30% of the full therapeutic dose) for 15 minutes per session, also one week before and one week after surgery. This procedure mimicked LLLT without providing therapeutic light exposure. Postoperative care and clinical assessments were identical to the LLLT group. Of the 30 patients initially assigned to the Control group, 13 were lost at the follow up leaving 17 patients (34 eyes) for the final analysis.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Low-Level Light Therapy — The intervention consists of non-invasive periocular photobiomodulation using the Eye-light® device (Espansione Marketing S.p.A., Italy), which delivers low-level monochromatic red light (633 ± 10 nm) through a specially designed mask. Participants receive two 15-minute sessions, one 7 days before and one 7 days after femtosecond laser-assisted in situ keratomileusis (Femto-LASIK). The treatment is designed to stimulate meibomian gland activity, improve tear film stability, and reduce ocular surface inflammation. This protocol is unique compared to standard post-refractive surgery care because it targets cellular mitochondrial activity to enhance tissue repair and anti-inflammatory effects. It is non-pharmacological, non-contact, and well-tolerated, making it suitable for perioperative application. The light is delivered through closed eyelids, ensuring safety and comfort, and the device used is CE-marked for ophthalmic applications.
  Arms: LLLT Group
Device: Sham (No Treatment) — Participants in the Control group underwent the same procedural setup as the LLLT group, using the Eye-light® device (Espansione Marketing S.p.A., Italy). Instead of delivering therapeutic light energy, the device operated in demo mode, emitting less than 30% of the full treatment power. This configuration mimicked the visual and sensory aspects of a low-level light therapy session without producing biologically effective photobiomodulation. Sham treatment consisted of two 15-minute sessions, one 7 days before and one 7 days after Femto-LASIK. This design ensured masking of participants and investigators while preventing active therapeutic exposure in the control group.
  Arms: Sham Group

SUMMARY:
This study evaluates the role of perioperative low-level light therapy (LLLT) in reducing dry eye disease (DED) symptoms after femtosecond laser-assisted in situ keratomileusis (Femto-LASIK). DED is one of the most frequent complications following Femto-LASIK, potentially affecting both visual recovery and patient satisfaction.

In this prospective, multicenter, randomized, double-masked, sham-controlled trial, adult patients undergoing Femto-LASIK were assigned to receive either periocular LLLT (Eye-light® )or sham treatment before and after surgery. Tear film parameters and ocular surface symptoms were assessed at baseline, 1 week, 1 month, and 3 months postoperatively.

Results showed that patients treated with LLLT maintained stable tear volume and reported fewer ocular discomfort symptoms compared with controls, who experienced significant declines. No adverse events related to LLLT were observed.

These findings suggest that perioperative LLLT is a safe and well-tolerated approach that may help preserve tear film stability and improve postoperative comfort in Femto-LASIK patients.

DETAILED DESCRIPTION:
This multicenter, randomized, double-masked, sham-controlled clinical trial was conducted to evaluate the efficacy and safety of perioperative low-level light therapy (LLLT) in preventing dry eye disease (DED) symptoms in patients undergoing femtosecond laser-assisted in situ keratomileusis (Femto-LASIK). The study was performed between August 2024 and June 2025 at the Centro Vista Eye Clinic and the Cai Ferate Clinical Hospital (Iași, Romania) in accordance with the Declaration of Helsinki and institutional ethics approval.

Dry eye disease is a multifactorial condition characterized by tear film instability, ocular surface inflammation, and neurosensory abnormalities. It is among the most common complications after corneal refractive surgery, largely due to the transection of corneal nerves during flap creation and excimer laser ablation, which disrupts the lacrimal functional unit and reduces tear production. This can impair visual recovery and reduce patient satisfaction.

LLLT is a non-invasive photobiomodulation technique that delivers low-intensity, monochromatic red light (633 ± 10 nm) to periocular tissues. It has been shown to improve mitochondrial function, modulate inflammatory pathways, and enhance meibomian gland activity, with potential benefits in ocular surface disease. Its role in the perioperative management of DED after LASIK, however, has not been fully explored.

Eligible participants were consecutive adults (≥18 years) scheduled for Femto-LASIK. Exclusion criteria included pre-existing ocular surface disease or DED, prior ocular surgery, autoimmune disease, use of systemic medications associated with DED, and any intraoperative or postoperative complications that could interfere with evaluation. Both eyes of each patient were included in the analysis.

Participants were randomized (1:1) to receive either LLLT or sham treatment. LLLT was administered with the Eye-light® device (Espansione Marketing S.p.A., Italy) for 15 minutes one week before and one week after surgery. Sham-treated patients underwent the same procedure with less than 30% of the treatment power, ensuring masking. All surgeries were performed by experienced surgeons using standardized LASIK techniques under topical anesthesia, followed by a uniform postoperative regimen including topical antibiotics, corticosteroids, and preservative-free artificial tears.

Clinical assessments were performed at baseline (T0), 1 week postoperatively (T1), 1 month (T2), and 3 months (T3).

Parameters included:

Non-invasive tear break-up time (NIBUT) Tear meniscus height (TMH) Lipid layer interferometry Schirmer I test Dry Eye Questionnaire-5 (DEQ-5)

The primary outcome was the preservation of tear volume and ocular surface parameters at 3 months postoperatively. Secondary outcomes included changes in patient-reported symptoms and tear film stability. Safety was evaluated by monitoring treatment-related adverse events and tolerability.

Statistical analysis was conducted using SPSS (version 30.0). Non-parametric and parametric tests were applied as appropriate, with p < 0.05 considered statistically significant. Sample size calculation ensured adequate power (>0.99) to detect clinically meaningful effects.

A total of 61 patients were randomized, of whom 40 (80 eyes) completed the study (23 in the LLLT group, 17 in the sham group). Patients receiving LLLT showed preserved tear meniscus height, stable Schirmer test values, and unchanged DEQ-5 scores over 3 months, whereas the sham group demonstrated significant deterioration in these parameters. No significant effects were found for NIBUT or interferometry. No treatment-related adverse events were reported, and LLLT was well tolerated.

This is the first prospective randomized trial to evaluate perioperative LLLT in Femto-LASIK patients. The results suggest that LLLT may protect ocular surface health, preserve tear volume, and improve patient comfort after refractive surgery. These findings support further research to optimize treatment protocols and confirm long-term benefits

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Scheduled for bilateral Femto-LASIK surgery for refractive error correction.
* Willing and able to provide written informed consent.
* Ability and willingness to comply with all study procedures and follow-up visits.
* Baseline ocular surface within normal limits (no pre-existing dry eye or ocular surface disease)

Exclusion Criteria:

* Prior diagnosis of ocular surface disease (OSD) or dry eye disease (DED).
* History of ocular surgery in either eye.
* Presence of ocular comorbidities such as glaucoma, corneal dystrophies, or active ocular infections.
* Current or regular use of topical ocular treatments, including lubricants, corticosteroids, cyclosporine, or other drugs for DED or OSD.
* Use of instrumental therapies for ocular surface or tear film optimization (e.g., thermal pulsation, IPL).
* Systemic treatments known to influence tear production (e.g., diuretics, antihistamines, antidepressants, hormone replacement therapy).
* Autoimmune diseases affecting the eyes, including Sjögren's syndrome or rheumatoid arthritis.
* Any intraoperative or postoperative complications that could interfere with ocular surface assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Preservation after Femto-LASIK with LLLT | Baseline (1 week preoperatively, T0) to 3 months postoperatively (T3)
  The Dry Eye Questionnaire-5 (DEQ-5) is a validated 5-item instrument used to assess the severity of subjective dry eye symptoms. The total score ranges from 0 to 22, with higher scores indicating greater symptom severity. The primary outcome is the change in total DEQ-5 score from baseline to 3 months after surgery, comparing the LLLT group to the control group.

SECONDARY OUTCOMES:
Non-Invasive Tear Break-Up Time (NIBUT) | Baseline (T0, 1 week preoperatively), 1 week postoperatively (T1), 1 month postoperatively (T2), 3 months postoperatively (T3)
  Non-Invasive Tear Break-Up Time (NIBUT) measures tear film stability by recording the interval (in seconds) between a complete blink and the first appearance of a dry spot on the corneal surface without fluorescein instillation. Higher NIBUT values indicate greater tear film stability, while lower values reflect more severe tear film instability. NIBUT will be assessed at baseline, 1 week, 1 month, and 3 months following treatment. The primary outcome is the change in NIBUT from baseline to 3 months postoperatively, comparing the LLLT and control groups.
Tear Lipid Layer Thickness (Interferometry) | Baseline (T0, 1 week preoperatively), 1 week postoperatively (T1), 1 month postoperatively (T2), 3 months postoperatively (T3)
  Tear Lipid Layer Thickness (LLT), assessed by interferometry, evaluates the quality and stability of the tear film lipid layer. Higher LLT values indicate a thicker lipid layer and greater tear film stability, while lower values reflect lipid deficiency and instability. LLT will be measured at baseline, 1 week, 1 month, and 3 months following treatment. The primary outcome is the change in LLT from baseline to 3 months postoperatively, comparing the LLLT and control groups.
Tear Meniscus Height (TMH) | Baseline (T0, 1 week preoperatively), 1 week postoperatively (T1), 1 month postoperatively (T2), 3 months postoperatively (T3)
  Tear Meniscus Height (TMH) is a non-invasive measure used to quantify tear volume by assessing the vertical height of the tear meniscus at the lower eyelid margin. Higher TMH values indicate greater tear volume, whereas lower values reflect aqueous deficiency. TMH will be evaluated at baseline, 1 week, 1 month, and 3 months following treatment. The primary outcome is the change in TMH from baseline to 3 months postoperatively, comparing the LLLT and control groups.
Schirmer Test (without anesthesia) | Baseline (T0, 1 week preoperatively), 1 week postoperatively (T1), 1 month postoperatively (T2), 3 months postoperatively (T3)
  The Schirmer test without anesthesia measures aqueous tear production by placing a standardized filter paper strip in the lower conjunctival fornix and recording the length of wetting (in millimeters) over 5 minutes. Higher values indicate greater tear secretion, while lower values reflect aqueous deficiency. The Schirmer test will be performed at baseline, 1 week, 1 month, and 3 months following treatment. The primary outcome is the change in Schirmer values from baseline to 3 months postoperatively, comparing the LLLT and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy "Grigore T. Popa" Iași,, Iași, Romania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including demographic information (age, sex), baseline and follow-up ocular surface parameters and treatment adherence data. No personally identifiable information will be disclosed. Data will be made available only upon reasonable request and for research purposes approved by an ethics committee or institutional review board.
Supporting Information: Study Protocol, SAP, CSR